CLINICAL TRIAL: NCT00457041
Title: Pilot Study Investigating Research Participants' Views on the Ethics of Clinical Research
Brief Title: Research Participants' Views on the Ethics of Clinical Research
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907073; 07-CC-N073
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-08

CONDITIONS: Rheumatic Diseases
Keywords: Trust; Decision Making; Vulnerability; Survey
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This pilot study will explore the usefulness of a series of questions asking about views of research from the perspective of minority and economically disadvantaged research participants. Racial and ethnic minorities are consistently under-represented in clinical research. This under-representation has been attributed primarily to an unwillingness to participate in research because of mistrust in the research establishment, especially in light of widely known historical examples of abuse. However, more recent data suggests that not being invited to participate in research, or stringent entry criteria, may contribute substantially to the low numbers of ethnic minority research participants. The perspectives of racial and ethnic minorities who are knowledgeable about or participating in research are important to understanding the kinds of vulnerabilities that exist and any important barriers to participation.

People 18 years of age and older from the Cardozo clinic in Washington, D.C., who are enrolled in the National Institute of Arthritis and Metabolic Studies' natural history study are eligible to participate in this protocol.

Participants are interviewed with questions about their own experiences in clinical research as well as some hypothetical research studies. Questions include participants' general views of clinical research, perceived risks and benefits of research, alternatives to research participation, the limits of what they would be willing to accept in research and types of research or research procedures they might perceive as unfair.

DETAILED DESCRIPTION:
In an effort to better understand ethical concerns about clinical research, this pilot study aims to explore the utility of a series of questions asking about views of research from the perspective of minority and economically disadvantaged research participants. Cognitive interviews will be conducted in English and Spanish with 10 participants of the NIAMS CHC at the Upper Cardozo Clinic in Washington DC. The interviewer will ask participants about their own experiences as well as some hypothetical research studies. Questionnaires will ask participants about their general views of the clinical research, perceived risks and benefits of research, alternatives to participation, the limits of what they would be willing to accept in research and types of research or research procedures they might perceive as unfair.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults (18 years and older) from Cardozo clinic who are enrolled in the NIAMS natural history study will be invited to participate in this interview study. The sample will include men and women who are primarily African American and Hispanic. Participants will be eligible if they are able and willing to give informed consent and can participate in an interview in English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01-17; Study Completion 2010-09-08

CONTACTS AND LOCATIONS:
Locations (1):
- NIAMS Community Health Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Shavers VL, Lynch CF, Burmeister LF. Factors that influence African-Americans' willingness to participate in medical research studies. Cancer. 2001 Jan 1;91(1 Suppl):233-6. doi: 10.1002/1097-0142(20010101)91:1+3.0.co;2-8. PMID 11148585
- [Background] Wendler D, Kington R, Madans J, Van Wye G, Christ-Schmidt H, Pratt LA, Brawley OW, Gross CP, Emanuel E. Are racial and ethnic minorities less willing to participate in health research? PLoS Med. 2006 Feb;3(2):e19. doi: 10.1371/journal.pmed.0030019. Epub 2005 Dec 6. PMID 16318411
- [Background] Gross CP, Filardo G, Mayne ST, Krumholz HM. The impact of socioeconomic status and race on trial participation for older women with breast cancer. Cancer. 2005 Feb 1;103(3):483-91. doi: 10.1002/cncr.20792. PMID 15597407